CLINICAL TRIAL: NCT05718752
Title: Characterization of the Metallome Fingerprint to Acute Intense Exercise: a Pilot Study on 40 Healthy Men and Women.
Brief Title: Characterization of the Plasma Metallomic Profile to Acute Exercise in Healthy Men and Women (METALEXO)
Acronym: METALEXO
Status: Completed | Type: Observational
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Frédéric Derbré, Associate Professor, University of Rennes 2
Other Study IDs: 2022-A02314-39
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Healthy Young Men; Healthy Young Women
Keywords: Maximal oxygen consumption; Physical performance; Metallomic profile; Iron metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Erythrocytes and plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy men: no intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: 30-min submaximal exercise test
- Healthy women: no intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: 30-min submaximal exercise test

INTERVENTIONS:
Diagnostic Test: Maximal incremental exercise test — Gas exchange are measured during all the test on ergocycle until oxygen consumption reach its maximum value
Diagnostic Test: 30-min submaximal exercise test — A 30-min submaximal test on ergocycle. Gas exchange are measured during all the test. Blood samples are collected before, at the end of exercise and after 3 hours of recovery

SUMMARY:
Among the various trace elements playing a key role in physical performance, iron is probably one of the most studied in the last 30 years. Iron is an essential component of both hemoglobin and myoglobin allowing an optimal oxygen delivery to organs, especially to skeletal muscle. Iron also plays a major role in the mitochondrial respiratory chain, as well as in the activity of numerous enzymes. Recent studies support the existence of a strong interaction between the iron metabolism and the other non-ferrous trace elements including among others zinc, copper or cobalt. The latter, but also other trace element metals could thus play an important role in physical performance. The finality of this project is thus 1) to determine the variations of plasma iron and non-ferrous metals in response to an acute exercise, 2) better understand the interactions between all these metals, 3) to determine if such responses to exercise are different or not depending on sex.

DETAILED DESCRIPTION:
Numerous trace element metals play an essential role in energy metabolism including magnesium, zinc or manganese (Heffernan et al., 2019). Elite men and women athletes with high energy demands consequently needs to compensate with food or drink intakes the lost and/or body misdistribution of these trace element metals during physical exercise. Trace element metals and their interactions in metabolic processes can play an important role in physical performance. However, the modulation of their plasma availability in response to acute exercise remains poorly understood (Heffernan et al., 2019). The Inductively Coupled Plasma Mass Spectrometry (ICP-MS) constitutes an efficient technology to detect and quantify all trace element metals in plasma and erythrocytes to answer this question.

Among the different trace element metals, iron is one of the most studied during the last 30 years. Iron is indeed an essential component of hemoglobin and myoglobin allowing an optimal oxygen delivery to organs, especially to skeletal muscle under contraction. Iron also plays a major role in the mitochondrial respiratory chain, as well as in the activity of numerous enzymes. Iron deficiency, especially in plasma iron availability, exerts deleterious consequences on sport performance by promoting iron deficiency anemia. Endurance athletes frequently exhibit iron deficiency (Sim et al., 2019), but the latter could also impact non-athletic populations, especially women (Mota et al., 2019). Disorders in iron metabolism during intense exercise could depend on several factors including hyperhecpidinemia (Roecker et al., 2005). High plasma hepcidin levels indeed contributes to reduction in plasma iron availability classically observed in elite athletes. Moreover, intravascular hemolysis combined to urinary, gastro-intestinal and/or sweat iron lost, could be also observed during prolonged intense exercise (Peeling et al., 2017). All together, these factors can directly impact functional capacities during physical exercise. Interestingly, recent studies support the existence of a strong interaction between the iron metabolism and the other non-ferrous trace elements including among others zinc, copper or cobalt (Loréal et al., 2014; Cavey et al., 2015). During intense physical exercise, the non-ferrous metals could thus directly or indirectly play a role in the modulation of iron import, storage or export in various kind of cells, and so functional capacities.

In this context, the pilot clinical study aims to characterize the plasma metallomic profile in response to an acute intense exercise in healthy men and women. All the volunteers (n=40) will perform 3 visits in the M2S lab: 1) an inclusion visit including anthropometric measures, dietary and physical activity surveys, 2) a second visit to perform the incremental cycling test, 3) a last visit to perform metabolic measures during a 30-min intense exercise (i.e. 90% of mechanical power at anaerobic threshold). Blood samples will be collected before, at the end of this intense exercise, and after 3 hours of recovery to determine in plasma systemic iron metabolism parameters and the concentrations of 29 non-ferrous metals.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 25 kg/m²
* Non smoker
* 150-300 min of moderate physical activity or 75-150 min of intensive physical activity per week.
* Written informed consent

Exclusion Criteria:

* Iron metabolism disorders (i.e. genetic hemochromatosis, thalassemia, anemia)
* Cardiovascular risks
* Metabolic diseases (e.g.diabetes)
* Use of non-steroidal anti-inflammatory drugs or aspirin
* Simultaneous participation in another research involving the human person or having recently participated in another research for which the exclusion period has not been completed.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physically active men and women
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Plasma iron availability | Week 3
  Serum iron levels and transferrin saturation will be determined before, just after the 30-min continuous ergocycle test and after 3 hours of recovery

SECONDARY OUTCOMES:
Plasma non-ferrous metals levels | Week 3
  Plasma concentrations of 29 non-ferrous metals will be determined before, just after the 30-min continuous ergocycle test and after 3 hours of recovery. Measurements will be performed using Inductively Coupled Plasma Mass Spectrometry (ICP/MS). A heat map will be performed to compare the hierarchical cluster analysis of plasma non-ferrous metals concentrations before and after physical exercise.
Plasma metallome fingerprint | Week 3
  Univariate linear regression will be determined to explore interactions between plasma concentrations of iron and non-ferrous metals.
Erythrocyte non-ferrous metals levels | Week 3
  Erythrocyte concentrations of 29 non-ferrous metals will be determined before, just after the 30-min continuous ergocycle test and after 3 hours of recovery. Measurements will be performed using Inductively Coupled Plasma Mass Spectrometry (ICP/MS).
Erythrocyte metallome fingerprint | Week 3
  Univariate linear regression will be determined to explore interactions between erythrocyte concentrations of iron and non-ferrous metals.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DERBRE, PhD, Principal Investigator — Laboratory of Movement, Sport and health Sciences (M2S)
Locations (1):
- University Rennes 2 - Laboratory "Movement, Sport and health Sciences", Bruz, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cleland CL, Hunter RF, Kee F, Cupples ME, Sallis JF, Tully MA. Validity of the global physical activity questionnaire (GPAQ) in assessing levels and change in moderate-vigorous physical activity and sedentary behaviour. BMC Public Health. 2014 Dec 10;14:1255. doi: 10.1186/1471-2458-14-1255. PMID 25492375
- [Background] Peeling P, McKay AKA, Pyne DB, Guelfi KJ, McCormick RH, Laarakkers CM, Swinkels DW, Garvican-Lewis LA, Ross MLR, Sharma AP, Leckey JJ, Burke LM. Factors influencing the post-exercise hepcidin-25 response in elite athletes. Eur J Appl Physiol. 2017 Jun;117(6):1233-1239. doi: 10.1007/s00421-017-3611-3. Epub 2017 Apr 13. PMID 28409396
- [Background] Heffernan SM, Horner K, De Vito G, Conway GE. The Role of Mineral and Trace Element Supplementation in Exercise and Athletic Performance: A Systematic Review. Nutrients. 2019 Mar 24;11(3):696. doi: 10.3390/nu11030696. PMID 30909645
- [Background] Roecker L, Meier-Buttermilch R, Brechtel L, Nemeth E, Ganz T. Iron-regulatory protein hepcidin is increased in female athletes after a marathon. Eur J Appl Physiol. 2005 Dec;95(5-6):569-71. doi: 10.1007/s00421-005-0055-y. Epub 2005 Oct 26. PMID 16249921
- [Background] Sim M, Garvican-Lewis LA, Cox GR, Govus A, McKay AKA, Stellingwerff T, Peeling P. Iron considerations for the athlete: a narrative review. Eur J Appl Physiol. 2019 Jul;119(7):1463-1478. doi: 10.1007/s00421-019-04157-y. Epub 2019 May 4. PMID 31055680
- [Background] Mota JO, Tounian P, Guillou S, Pierre F, Membre JM. Estimation of the Burden of Iron Deficiency Anemia in France from Iron Intake: Methodological Approach. Nutrients. 2019 Sep 1;11(9):2045. doi: 10.3390/nu11092045. PMID 31480641
- [Background] Loreal O, Cavey T, Bardou-Jacquet E, Guggenbuhl P, Ropert M, Brissot P. Iron, hepcidin, and the metal connection. Front Pharmacol. 2014 Jun 4;5:128. doi: 10.3389/fphar.2014.00128. eCollection 2014. PMID 24926268
- [Background] Cavey T, Ropert M, de Tayrac M, Bardou-Jacquet E, Island ML, Leroyer P, Bendavid C, Brissot P, Loreal O. Mouse genetic background impacts both on iron and non-iron metals parameters and on their relationships. Biometals. 2015 Aug;28(4):733-43. doi: 10.1007/s10534-015-9862-8. Epub 2015 Jun 4. PMID 26041486